CLINICAL TRIAL: NCT01983345
Title: Prenatal Surgical Repair of Fetal Myelomeningocele
Acronym: PRIUM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P121103; 2013-A00385-40 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2013-11-07; First posted 2013-11-14 (Estimated); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Foetus With Myelomeningocele
Keywords: Myelomeningocele; Arnold Chiari malformation; Spina bifida
MeSH Terms: conditions — Meningomyelocele; Arnold-Chiari Malformation; Spinal Dysraphism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): No prenatal surgical repair of myelomeningocele
- Case - open surgical repair (Experimental): Prenatal surgical repair of fetal myelomeningocele
  Interventions: Procedure: prenatal surgical repair of fetal myelomeningocele

INTERVENTIONS:
Procedure: prenatal surgical repair of fetal myelomeningocele — open surgical repair of myelomeningocele before 26 weeks gestational age
  Arms: Case - open surgical repair

SUMMARY:
The open surgical repair of myelomeningoceles before 26 weeks gestational age provides a correction of the anomaly of Chiarri, reduces the incidence of ventriculomegaly (defined as a measure of the ventricles at the crossroads ≥ 10 mm), and get a lower of injury than one corresponding to the anatomical defect (as defined by the last upper normal vertebra before the defect).

The purpose of this study is to introduce in France an innovative technique for prenatal repair of myelomeningocele until now developed only on the American continent.

DETAILED DESCRIPTION:
Spina bifida (SB) represents one of the most severe congenital malformation of the central nervous system and amenable to prenatal diagnosis. In the past 20 years, prenatal repair of SB has become an established technique.

The PRIUM study will include 10 cases of fetuses with prenatal diagnosis of SB and for whom the maternal willing will be to continue the pregnancy. A surgical prenatal repair of the defect will be planed at 19-25+6 weeks gestation following maternal laparotomy and hysterotomy under maternal general anesthesia. The delivery will be planed at 36 weeks'. Postnatal evaluation of the neonates will be scheduled at birth, 1 month, 12 months and 36 months of age. Those data will be matched to controls who have underwent a conventional postnatal repair of the SB

ELIGIBILITY:
Inclusion Criteria:

* patient of majority age, with an assumption by health insurance, understanding and speaking French
* A term between 19 and 25 +6 weeks gestational age (not for control)
* Single-Pregnancy
* Normal fetal karyotype
* Myelomeningocele with higher-level defect between S1 and T1
* Placenta not low-inserted or not covering
* Fault-isolated ultrasound reference

Exclusion Criteria:

* Age under 18 years
* Patient foreigner who understands not French
* Multiple Pregnancy
* Low Placenta inserted or covering
* Severe kyphosis
* Placental abruption
* Fetal malformation unrelated to the existence of myelomeningocele (the existence of a malposition of one or both feet do not represent an exclusion criterion)
* Increased risk of preterm birth: a history of preterm delivery before 37 weeks gestational age, cervical length <26 mm before 26 weeks gestational age (not for control)
* Bleeding active between 20 and 26 weeks gestational age (not for control)
* Maternal obesity with BMI> 35 (not for control)
* History of uterine surgery involving the anterior surface of the uterus (not for control)
* Maternal contradiction in surgery or general anesthesia (not for control)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2014-07-10 (Actual); Primary Completion 2021-07-28 (Actual); Study Completion 2021-07-28 (Actual)

PRIMARY OUTCOMES:
Arnold Chiari anomaly at birth | Day 0
  the existence of an Arnold Chiari anomaly at birth
Defect | 3 years
  the level difference between the observed level of injury and the anatomical level of the defect (as defined by the last normal upper vertebra before the defect)

CONTACTS AND LOCATIONS:
Overall Officials: Michel Zerah, MD, PhD, Study Director — Assistance Publique - Hôpitaux de Paris; Jean-Marie Jouannic, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hopital Armand Trousseau, APHP, Paris, PARIS, France

REFERENCES:
- [Background] Friszer S, Dhombres F, Di Rocco F, Rigouzzo A, Garel C, Guilbaud L, Forin V, Moutard ML, Zerah M, Jouannic JM. [Preliminary results from the French study on prenatal repair for fetal myelomeningoceles (the PRIUM study)]. J Gynecol Obstet Biol Reprod (Paris). 2016 Sep;45(7):738-44. doi: 10.1016/j.jgyn.2015.09.002. Epub 2015 Nov 10. French. PMID 26566108
- [Background] Guilbaud L, Maurice P, Lallemant P, De Saint-Denis T, Maisonneuve E, Dhombres F, Friszer S, Di Rocco F, Garel C, Moutard ML, Lachtar MA, Rigouzzo A, Forin V, Zerah M, Jouannic JM. Open fetal surgery for myelomeningocele repair in France. J Gynecol Obstet Hum Reprod. 2021 Nov;50(9):102155. doi: 10.1016/j.jogoh.2021.102155. Epub 2021 Apr 26. PMID 33915336